CLINICAL TRIAL: NCT02171156
Title: Multi-center Open-label Expanded Access Program of Oral Nintedanib 150 mg Twice Daily in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Expanded Access Program of Nintedanib in Patients With Idiopathic Pulmonary Fibrosis (EAP)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199.177
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: nintedanib — soft gelatin capsule

SUMMARY:
To provide early access and to evaluate the safety and tolerability of nintedanib in patients with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion criteria:

1. Signed Informed Consent consistent with ICH-GCP and local laws signed prior to entry into the trial;
2. Male or female patients aged >=40 years at Visit 1;
3. IPF diagnosis based upon the American Thoracic Society (ATS)/European Respiratory Society (ERS) /Japanese Respiratory Society (JRS)/Latin American Thoracic Society (ALAT) IPF 2011 guideline within 5 years of visit 1;
4. Carbon monoxide diffusing capacity (DLCO)(corrected for Haemoglobin (Hb)): 30%-79% predicted of normal, per institutional standards at the clinic site, at Visit 1;
5. Forced Vital Capacity (FVC) >= 50% predicted of normal, per institutional standards at the clinic site, at Visit 1.

Exclusion criteria:

1. Eligible to participate or participating in an ongoing actively accruing clinical trial with nintedanib in the treatment of IPF.

   Laboratory parameters from Visit 1 must satisfy entry criteria as shown below. Abnormal laboratory parameters may be re-tested if a measurement error is suspected (e.g., there was no abnormal result of this test in the recent history of the patient and there is no related clinical sign). The results of the re-test should be reported within the Screening period (i.e., 28 days of signing the informed consent form).
2. ALT, AST > 1.5 times upper limit of normal (ULN);
3. Total Bilirubin > 1.5 times upper limit of normal (ULN);
4. Bleeding risk:

   1. patients who require: fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, dabigatran, heparin, hirudin, etc.), or high-dose antiplatelet therapy. Exceptions: prophylactic low dose heparin or heparin flush as needed for maintenance of an indwelling intravenous device (e.g., enoxaparin 4000 IU s.c. per day) and prophylactic use of antiplatelet therapy (e.g., acetylsalicylic acid up to 325 mg/d, or clopidogrel at 75 mg/d, or equivalent doses of other antiplatelet therapy);
   2. history of hemorrhagic central nervous system (CNS) event within 12 months of Visit 1;
   3. any of the following within 3 months of Visit 1;

      * hemoptysis or haematuria
      * active gastro-intestinal bleeding or ulcers
      * major injury or surgery
   4. coagulation parameters:

      * international normalised ratio (INR) > 2
      * prothrombin time (PT) and partial thromboplastin time (PTT) > 150% of institutional upper limit of normal (ULN)
5. Planned major surgery within the next 3 months, including lung transplantation, major abdominal or major intestinal surgery;
6. Thrombotic risk:

   1. known inherited predisposition to thrombosis
   2. history of thrombotic event (including stroke and transient ischemic attacks) within 12 months of Visit 1;
7. Cardiac disease:

   1. Myocardial infarction within 6 months of Visit 1
   2. Unstable angina within 1 month of Visit 1;
8. Current or planned usage (during the course of this trial) of any other investigational drug during the course of this trial;
9. Current or planned treatment (during the course of this trial) with: pirfenidone, azathioprine, cyclophosphamide, cyclosporine, prednisone >15 mg daily or > 30 mg every 2 days OR equivalent dose of other oral corticosteroids, as well as those listed in exclusion criteria #4 (bleeding risk);
10. Permanent discontinuation of nintedanib within a clinical trial, due to adverse events considered drug-related;
11. Known hypersensitivity to nintedanib or its excipients;
12. A disease or condition which in the opinion of treating physician may put the patient at risk because of participation in this trial or limit the patient's ability to participate in this trial;
13. Alcohol or drug abuse which in the opinion of the treating physician would interfere with participation;
14. Women (of child-bearing potential) who are unwilling to use acceptable methods of contraception;
15. Pregnancy or breast feeding (female patients must have a negative pregnancy test (ß-HCG test in urine or serum) prior to commencing trial treatment).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- United States (7):
  - 1199.177.1003 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1199.177.1012 Boehringer Ingelheim Investigational Site, Skokie, Illinois
  - 1199.177.1014 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 1199.177.1002 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1199.177.1011 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1199.177.1022 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1199.177.1067 Boehringer Ingelheim Investigational Site, Houston, Texas